CLINICAL TRIAL: NCT06870916
Title: Supporting Informed Decision Making About Multi-cancer Early Detection Testing
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1925; NCI-2025-01726 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Multi-cancer Early Detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multi-cancer Early Detection: Participants will participate in a focus group discussion asking about participants knowledge, preferences, and concerns for MCEDs. During the focus group discussion, investigators will specifically talk about what the tests are and how to decide to get the test as well as their risks and benefits.
  Interventions: Other: Multi-cancer Early Detection

INTERVENTIONS:
Other: Multi-cancer Early Detection — Participants will participate in a focus group discussion asking about your knowledge, preferences, and concerns for MCEDs. During the focus group discussion, investigators will specifically talk about what the tests are and how to decide to get the test as well as their risks and benefits.

SUMMARY:
To develop a new participant educational aid that can be used by participants to support informed decision-making about Multi-Cancer Early Detection (MCED) tests, which are new blood-based screening tests.

DETAILED DESCRIPTION:
To develop a prototype participant educational aid that can be used by participants to support informed decision making about MCED testing. The aims of the pilot project include the following:

1. Conduct focus groups to explore preferences and concerns about MCED testing among adults of screening age.
2. Based on salient themes from focus group discussion, develop and administer surveys to explore preferences and concerns about MCED testing among adults of screening age.
3. Using findings from the focus groups and surveys, develop prototype patient educational aids about MCED testing following a user-centered design strategy.

ELIGIBILITY:
Inclusion Criteria:

• Recruitment and eligibility will be assessed by CCETR.CCETR staff will help distribute recruitment flyers, assess subject eligibility, and refer eligible subjects to the research team (Appendix B, C & I).

Exclusion Criteria:

• History of cancer other than basil cell and squamous cell skin cancer, per self-report.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Volk, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org